CLINICAL TRIAL: NCT00419185
Title: Internal Limiting Membrane (ILM)- Peeling With Indocyanine Green or Trypan Blue in Macular Hole Surgery: A Prospective Randomized Trial
Brief Title: Indocyanine Green or Trypan Blue for Delamination of the Internal Limiting Membrane in Macular Hole Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKSH
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2007-01-08 (Estimated); Status verified 2007-01

CONDITIONS: Idiopathic Macular Hole
Keywords: macular hole surgery; indocyanine green; trypan blue; internal limiting membrane

INTERVENTIONS:
Procedure: Delamination of the Internal limiting membrane

SUMMARY:
To evaluate the anatomical and visual outcomes after vitrectomy and internal limiting membrane (ILM) peeling with indocyanine green (ICG) or trypan blue (TB) for idiopathic macular hole repair in a prospective randomized trial.

DETAILED DESCRIPTION:
In several clinical trials the positive effect of inner limiting membrane peeling (ILM) on anatomical and functional outcome in macular hole surgery has been reported. Controversies, however, exist regarding the application and possible toxicity of dyes, facilitating the surgical procedure. Since dyes were introduced for ILM peeling several authors reported on the use of indocyanine green and trypan blue (TB) for membrane peeling or ILM removal. Recent experimental and clinical reports raise concern about the safety of ICG-assisted membrane peeling. Morphological and functional damage was described in an animal model, in human donor eyes, in cultured human pigment epithelial cells and in clinical studies using ICG in macular surgery. The intraocular tolerance of TB has been demonstrated in rabbit eyes and in retinal pigment epithelium cell viability studies. Higher concentrations of TB (0.6 or 4 mg/ml) lead to toxicity on cultured RPE cells, but the application of lower clinically relevant levels did not show any significant effect. A recent retrospective comparative analysis indicates that TB may be the safer dye. They found better anatomical and functional results than with the use of ICG.

Therefore, the aim of this study was to compare the anatomical and functional outcome after dye-assisted peeling of the ILM in patients with idiopathic macular holes using ICG or TB in a prospective and randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic macular holes stage II-IV according to the classification proposed by Gass and a visual acuity of at least 20/200 entered this study.

Exclusion Criteria:

* Patients with secondary macular holes, previous intraocular surgery, except for uneventful cataract extraction and patients with ocular disorders that might interfere with vision such as severe cataract, exudative age-related macular degeneration or diabetic retinopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-04; Study Completion 2005-01

PRIMARY OUTCOMES:
Primary outcome was ETDRS visual acuity (VA: snellen equivalent) at two meters 3 months after surgery.
Assignment to ICG or TB dye was performed by the Institute of Medical Biometry and Statistics of the University Luebeck per telephone immediately before surgery. Allocation to treatment arms was done with a permuted block randomization with block size 20

SECONDARY OUTCOMES:
Secondary outcome measures were successful hole closure defined only as complete closure of the inner retinal dehiscence determined by OCT,
cystoid macular edema as revealed by fluorescein angiography (FLA) and
postoperative scotoma shown by SLO-microperimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Hans M Hoerauf, Prof., Principal Investigator — Eye Clinic, University Schleswig Holstein, Campus Lübeck
Locations (1):
- Eye Clinic, University Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Kadonosono K, Itoh N, Uchio E, Nakamura S, Ohno S. Staining of internal limiting membrane in macular hole surgery. Arch Ophthalmol. 2000 Aug;118(8):1116-8. doi: 10.1001/archopht.118.8.1116. PMID 10922208
- [Background] Brooks HL Jr. Macular hole surgery with and without internal limiting membrane peeling. Ophthalmology. 2000 Oct;107(10):1939-48; discussion 1948-9. doi: 10.1016/s0161-6420(00)00331-6. PMID 11013203
- [Background] Haritoglou C, Gass CA, Schaumberger M, Gandorfer A, Ulbig MW, Kampik A. Long-term follow-up after macular hole surgery with internal limiting membrane peeling. Am J Ophthalmol. 2002 Nov;134(5):661-6. doi: 10.1016/s0002-9394(02)01751-8. PMID 12429240
- [Background] Kuhn F. Point: to peel or not to peel, that is the question. Ophthalmology. 2002 Jan;109(1):9-11. doi: 10.1016/s0161-6420(01)00992-7. No abstract available. PMID 11772571
- [Background] Burk SE, Da Mata AP, Snyder ME, Rosa RH Jr, Foster RE. Indocyanine green-assisted peeling of the retinal internal limiting membrane. Ophthalmology. 2000 Nov;107(11):2010-4. doi: 10.1016/s0161-6420(00)00375-4. PMID 11054324
- [Background] Li K, Wong D, Hiscott P, Stanga P, Groenewald C, McGalliard J. Trypan blue staining of internal limiting membrane and epiretinal membrane during vitrectomy: visual results and histopathological findings. Br J Ophthalmol. 2003 Feb;87(2):216-9. doi: 10.1136/bjo.87.2.216. PMID 12543755
- [Background] Enaida H, Sakamoto T, Hisatomi T, Goto Y, Ishibashi T. Morphological and functional damage of the retina caused by intravitreous indocyanine green in rat eyes. Graefes Arch Clin Exp Ophthalmol. 2002 Mar;240(3):209-13. doi: 10.1007/s00417-002-0433-7. Epub 2002 Feb 15. PMID 11935278
- [Background] Gandorfer A, Haritoglou C, Gandorfer A, Kampik A. Retinal damage from indocyanine green in experimental macular surgery. Invest Ophthalmol Vis Sci. 2003 Jan;44(1):316-23. doi: 10.1167/iovs.02-0545. PMID 12506091
- [Background] Sippy BD, Engelbrecht NE, Hubbard GB, Moriarty SE, Jiang S, Aaberg TM Jr, Aaberg TM Sr, Grossniklaus HE, Sternberg P Jr. Indocyanine green effect on cultured human retinal pigment epithelial cells: implication for macular hole surgery. Am J Ophthalmol. 2001 Sep;132(3):433-5. doi: 10.1016/s0002-9394(01)01061-3. PMID 11530072
- [Background] Stalmans P, Van Aken EH, Veckeneer M, Feron EJ, Stalmans I. Toxic effect of indocyanine green on retinal pigment epithelium related to osmotic effects of the solvent. Am J Ophthalmol. 2002 Aug;134(2):282-5. doi: 10.1016/s0002-9394(02)01468-x. PMID 12140045
- [Background] Engelbrecht NE, Freeman J, Sternberg P Jr, Aaberg TM Sr, Aaberg TM Jr, Martin DF, Sippy BD. Retinal pigment epithelial changes after macular hole surgery with indocyanine green-assisted internal limiting membrane peeling. Am J Ophthalmol. 2002 Jan;133(1):89-94. doi: 10.1016/s0002-9394(01)01293-4. PMID 11755843
- [Background] Wolf S, Reichel MB, Wiedemann P, Schnurrbusch UEK. Clinical findings in macular hole surgery with indocyanine green-assisted peeling of the internal limiting membrane. Graefes Arch Clin Exp Ophthalmol. 2003 Jul;241(7):589-592. doi: 10.1007/s00417-003-0673-1. Epub 2003 May 8. PMID 12736727
- [Background] Ando F, Yasui O, Hirose H, Ohba N. Optic nerve atrophy after vitrectomy with indocyanine green-assisted internal limiting membrane peeling in diffuse diabetic macular edema. Adverse effect of ICG-assisted ILM peeling. Graefes Arch Clin Exp Ophthalmol. 2004 Dec;242(12):995-9. doi: 10.1007/s00417-004-0864-4. Epub 2004 Jul 17. PMID 15592868
- [Background] Gass CA, Haritoglou C, Schaumberger M, Kampik A. Functional outcome of macular hole surgery with and without indocyanine green-assisted peeling of the internal limiting membrane. Graefes Arch Clin Exp Ophthalmol. 2003 Sep;241(9):716-20. doi: 10.1007/s00417-003-0710-0. Epub 2003 Aug 13. PMID 12920526
- [Background] Kwok AK, Yeung CK, Lai TY, Chan KP, Pang CP. Effects of trypan blue on cell viability and gene expression in human retinal pigment epithelial cells. Br J Ophthalmol. 2004 Dec;88(12):1590-4. doi: 10.1136/bjo.2004.044537. PMID 15548818
- [Background] Lee KL, Dean S, Guest S. A comparison of outcomes after indocyanine green and trypan blue assisted internal limiting membrane peeling during macular hole surgery. Br J Ophthalmol. 2005 Apr;89(4):420-4. doi: 10.1136/bjo.2004.049684. PMID 15774917
- [Background] Horio N, Horiguchi M. Effect on visual outcome after macular hole surgery when staining the internal limiting membrane with indocyanine green dye. Arch Ophthalmol. 2004 Jul;122(7):992-6. doi: 10.1001/archopht.122.7.992. PMID 15249363
- [Background] Da Mata AP, Burk SE, Riemann CD, Rosa RH Jr, Snyder ME, Petersen MR, Foster RE. Indocyanine green-assisted peeling of the retinal internal limiting membrane during vitrectomy surgery for macular hole repair. Ophthalmology. 2001 Jul;108(7):1187-92. doi: 10.1016/s0161-6420(01)00593-0. PMID 11425673
- [Background] Kwok AK, Lai TY, Yuen KS, Tam BS, Wong VW. Macular hole surgery with or without indocyanine green stained internal limiting membrane peeling. Clin Exp Ophthalmol. 2003 Dec;31(6):470-5. doi: 10.1046/j.1442-9071.2003.00709.x. PMID 14641152
- [Background] Ando F, Sasano K, Ohba N, Hirose H, Yasui O. Anatomic and visual outcomes after indocyanine green-assisted peeling of the retinal internal limiting membrane in idiopathic macular hole surgery. Am J Ophthalmol. 2004 Apr;137(4):609-14. doi: 10.1016/j.ajo.2003.08.038. PMID 15059697
- [Background] Lochhead J, Jones E, Chui D, Lake S, Karia N, Patel CK, Rosen P. Outcome of ICG-assisted ILM peel in macular hole surgery. Eye (Lond). 2004 Aug;18(8):804-8. doi: 10.1038/sj.eye.6701328. PMID 14752502
- [Background] Slaughter K, Lee IL. Macular hole surgery with and without indocyanine green assistance. Eye (Lond). 2004 Apr;18(4):376-8. doi: 10.1038/sj.eye.6700666. PMID 15069433
- [Background] Haritoglou C, Gass CA, Schaumberger M, Ehrt O, Gandorfer A, Kampik A. Macular changes after peeling of the internal limiting membrane in macular hole surgery. Am J Ophthalmol. 2001 Sep;132(3):363-8. doi: 10.1016/s0002-9394(01)01093-5. PMID 11530049
- [Background] Paques M, Genevois O, Regnier A, Tadayoni R, Sercombe R, Gaudric A, Vicaut E. Axon-tracing properties of indocyanine green. Arch Ophthalmol. 2003 Mar;121(3):367-70. doi: 10.1001/archopht.121.3.367. PMID 12617707
- [Background] Uemoto R, Yamamoto S, Takeuchi S. Changes in retinal pigment epithelium after indocyanine green-assisted internal limiting lamina peeling during macular hole surgery. Am J Ophthalmol. 2005 Oct;140(4):752-5. doi: 10.1016/j.ajo.2005.04.035. PMID 16226539
- [Background] Haritoglou C, Gandorfer A, Schaumberger M, Tadayoni R, Gandorfer A, Kampik A. Light-absorbing properties and osmolarity of indocyanine-green depending on concentration and solvent medium. Invest Ophthalmol Vis Sci. 2003 Jun;44(6):2722-9. doi: 10.1167/iovs.02-1283. PMID 12766079
- [Background] Rezai KA, Farrokh-Siar L, Gasyna EM, Ernest JT. Trypan blue induces apoptosis in human retinal pigment epithelial cells. Am J Ophthalmol. 2004 Sep;138(3):492-5. doi: 10.1016/j.ajo.2004.03.033. PMID 15364242
- [Background] Jackson TL, Hillenkamp J, Knight BC, Zhang JJ, Thomas D, Stanford MR, Marshall J. Safety testing of indocyanine green and trypan blue using retinal pigment epithelium and glial cell cultures. Invest Ophthalmol Vis Sci. 2004 Aug;45(8):2778-85. doi: 10.1167/iovs.04-0320. PMID 15277504
- [Background] Gale JS, Proulx AA, Gonder JR, Mao AJ, Hutnik CM. Comparison of the in vitro toxicity of indocyanine green to that of trypan blue in human retinal pigment epithelium cell cultures. Am J Ophthalmol. 2004 Jul;138(1):64-9. doi: 10.1016/j.ajo.2004.02.061. PMID 15234283
- [Background] Kwok AK, Lai TY, Yew DT, Li WW. Internal limiting membrane staining with various concentrations of indocyanine green dye under air in macular surgeries. Am J Ophthalmol. 2003 Aug;136(2):223-30. doi: 10.1016/s0002-9394(02)02144-x. PMID 12888042
- [Derived] Beutel J, Dahmen G, Ziegler A, Hoerauf H. Internal limiting membrane peeling with indocyanine green or trypan blue in macular hole surgery: a randomized trial. Arch Ophthalmol. 2007 Mar;125(3):326-32. doi: 10.1001/archopht.125.3.326. PMID 17353402